CLINICAL TRIAL: NCT02774824
Title: A 9-month Extension Study to: A Study to Evaluate the Use of SOMVC001 (GALA) Vascular Conduit Preservation Solution in Patients Undergoing Coronary Artery Bypass Grafting (CABG)
Brief Title: 9 Months Extension Study of SOMVC001 Study (GALA) Vascular Conduit Preservation Solution
Status: Completed | Type: Observational
Sponsor: Perrault Louis P. (Other)
Collaborators: Montreal Heart Institute (Other); Somahlution LLC (Industry)
Responsible Party: Sponsor-Investigator, Perrault Louis P., Cardiovascular Thoracic Surgeon, Montreal Heart Institute
Organization: Montreal Heart Institute (Other)
Other Study IDs: 003-10
Record Dates: First submitted 2016-05-05; First posted 2016-05-17 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CABG patients from protocol 003-03: Patients who will agree to be followed for an additional 9 months, which include:
  2 phone calls at 6 and 9 months after coronary artery bypass graft surgery
  1 clinic visit at 12 months after coronary artery bypass graft surgery ( 64-slice or better MDCT angiography)

SUMMARY:
This is a 9-months extension to the following study, protocol number: 003-03: "A study to evaluate the use of SOMVC001 (GALA) vascular conduit preservation solution in patients undergoing coronary artery bypass grafting (GABG)". Participation is allowed exclusively to participants enrolled in the main protocol SOMVC001 (GALA).

DETAILED DESCRIPTION:
Patients enrolled in this 9-months extension study of SOMVC001 (GALA) will be contacted by phone twice: 6 months and 9 months after a coronary artery bypass graft (CABG) surgery. During these phone call visits and at twelve months post CABG surgery, adverse events and/or concomitant medication changes will be collected from the participant. Twelve months after the CABG surgery procedure, imaging will be performed using 64-slice or better MDCT-scan angiography. The study participation ends at this MDCT-scan visit.

In detail, will be recorded incidence of composite safety outcomes consisting of Major Adverse Cardiac Events (MACE) (death, myocardial infarction [MI], and repeat revascularization), angina, arrhythmias, shortness of breath [SOB], decreased lumen change, graft occlusion and significant stenosis based on Fitzgibbon's scale B and O, following CABG surgery.

Patients in this study are their own control; they receive two SVG; one exposed to GALA and the other exposed to heparinized dose saline. The effect of treatment (GALA vs. Saline) will be evaluated on paired grafts within-person. Therefore, treatment effect will be presented by graft and not by patient. Only adverse clinical events will be presented by patient including their potential relationship to the study product.

ELIGIBILITY:
Inclusion Criteria:

* patients from protocol #003-03 who agree to be followed for an additional 9 months by signing informed consent.

Exclusion Criteria:

* patients who have a contraindication to undergo MDCT angiography ant 12 months post CABG surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had a coronary artery bypass graft surgery (CABG), and took part in previous main study of SOMVC001 (GALA) protocol ID # 003-03 .
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-08-24 (Actual); Study Completion 2017-08-24 (Actual)

PRIMARY OUTCOMES:
It will be measured and reported, the mean lumen diameter of paired grafts (one treated vs one not treated) within-person. Mean lumen diameter will be expressed in millimeter (mm) . | At twelve months following CABG surgery
  performing a 64-slice or better multi-detector computed tomography (MDCT) angiography, by assessing the magnitude of change in the mean lumen diameter of paired grafts within person, one year post- surgery.
It will be measured and reported, the maximum stenosis of paired grafts (one treated vs one not treated) within-person. The maximum stenosis will be expressed in millimeter (mm). | At twelve months following CABG surgery
  Performing a 64-slice or better multi-detector computed tomography (MDCT) angiography by assessing the magnitude of change at maximum stenosis of paired grafts within person, one year post-surgery.
The incidence of vein graft thrombosis will be measured as total graft occlusion | At twelve months following CABG surgery
  Using a 64-slice or better multi-detector computed tomography (MDCT) angiography.

SECONDARY OUTCOMES:
The change in maximal stenosis will be measured and expressed in millimeter (mm) as changes over time. | from 4-6 weeks to 12 months and from 3 months to 12 months following CABG surgery
  Using a 64-slice or better multi-detector computed tomography (MDCT) angiography.
The change in lumen will be measured and expressed in millimeter (mm) as changes over time. | from 4-6 weeks to 12 months and from 3 months to 12 months following CABG surgery.
  Using a 64-slice or better multi-detector computed tomography (MDCT) angiography.
The change in vessel diameter will be measured and expressed in millimeter (mm) as changes over time. | from 4-6 weeks to 12 months and from 3 months to 12 months following CABG surgery
  Using a 64-slice or better multi-detector computed tomography (MDCT) angiography.
The change in total wall thickness will be measured and expressed in millimeter (mm) as changes over time. | from 4-6 weeks to 12 months and from 3 months to 12 months following CABG surgery
  Using a 64-slice or better multi-detector computed tomography (MDCT) angiography.

CONTACTS AND LOCATIONS:
Overall Officials: Louis P Perrault, MD, PhD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ben Ali W, Voisine P, Olsen PS, Jeanmart H, Noiseux N, Goeken T, Satishchandran V, Cademartiri F, Cutter G, Veerasingam D, Brown C, Emmert MY, Perrault LP. DuraGraft vascular conduit preservation solution in patients undergoing coronary artery bypass grafting: rationale and design of a within-patient randomised multicentre trial. Open Heart. 2018 Apr 13;5(1):e000780. doi: 10.1136/openhrt-2018-000780. eCollection 2018. PMID 29682294